CLINICAL TRIAL: NCT00624221
Title: A Prospective, Randomized, Single Center Study Evaluating Use of Surgeon- and Eye Bank-prepared Donor Tissue for Descemet's Stripping and Endothelial Keratoplasty, a Type of Cornea Transplant
Brief Title: Study of Eye Bank Pre-cut Donor Grafts for Endothelial Keratoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornea Research Foundation of America (Other)
Collaborators: North Carolina Lion's Eye Bank (Unknown); Price Vision Group (Industry)
Responsible Party: Francis W. Price, Jr. MD, Cornea Research Foundation of America
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-10
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Results first posted 2010-03-12 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2010-10

CONDITIONS: Fuchs Endothelial Dystrophy; Corneal Edema
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Edema | interventions — Descemet Stripping Endothelial Keratoplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): An Eye bank pre-cut the donor grafts used for the corneal transplant procedures.
  Interventions: Procedure: Descemet's stripping endothelial keratoplasty
- 2 (Active Comparator): The surgeon dissected the donor grafts used for the transplant procedures.
  Interventions: Procedure: Descemet's stripping endothelial keratoplasty

INTERVENTIONS:
Procedure: Descemet's stripping endothelial keratoplasty — Small incision corneal transplant procedure to treat dysfunctional endothelium.

SUMMARY:
Descemet's stripping with endothelial keratoplasty (DSEK) is a cornea-sparing transplant technique that replaces only the diseased endothelial cell layer of the patient's cornea. The DSEK technique requires lamellar dissection of the donor tissue prior to implantation in the patient's eye. The surgeon usually dissects the donor cornea with a microkeratome at the time of surgery. Recently some eye banks have begun to pre-cut the donor graft as an added service. The purpose of this study was to compare outcomes with eye bank pre-cut and surgeon-dissected donor grafts for DSEK.

ELIGIBILITY:
Inclusion Criteria:

* candidate for Descemet's stripping with endothelial keratoplasty
* at least 21 years old
* willing and able to return for scheduled follow-up visits
* reads and signs Informed Consent document

Exclusion Criteria:

* visual acuity of less than 20/400 in fellow eye
* known sensitivity to planned study concomitant medications

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr, MD, Principal Investigator — Cornea Research Foundation of America
Locations (1):
- Cornea Research Foundation of America, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Eye Bank Pre-cut Grafts: An Eye bank pre-cut the donor grafts used for the corneal transplant procedures.
- Surgeon Dissected Grafts: The surgeon dissected the donor grafts used for the transplant procedures.
Period: Overall Study
Arm/Group | Eye Bank Pre-cut Grafts | Surgeon Dissected Grafts
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eye Bank Pre-cut Grafts | Surgeon Dissected Grafts | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (12) | 72 (13) | 71 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Cell Loss
Description: Endothelial cell density was measured by specular or confocal microscopy. Percent cell loss was calculated by subtracting the graft endothelial cell density measured at 6 months from the baseline donor endothelial cell density and dividing by the baseline donor endothelial cell density then multiplying by 100.
Time Frame: 6 months after grafting
Measure: Mean (Standard Deviation); unit: percentage of endothelial cell loss
Arm/Group | Eye Bank Pre-cut Grafts | Surgeon Dissected Grafts
Number analyzed (Participants) | 20 | 20
percentage of endothelial cell loss | 28 (20) | 36 (18)
Statistical Analysis 1: Comparison: Eye Bank Pre-cut Grafts vs Surgeon Dissected Grafts; Test type: Non-Inferiority or Equivalence — The sample size of 40 subjects was estimated based on having 80% power to determine greater than 10% difference in cell loss between groups with estimated standard deviation of 17 and estimated correlation of 0.5; p = 0.10, paired difference t-test

2. Secondary Outcome: Best Corrected Vision
Time Frame: 6 months and 1 year after grafting
Reporting Status: Not Posted

3. Secondary Outcome: Graft Dislocation
Time Frame: 1 day to 1 month after grafting
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Eye Bank Pre-cut Grafts | Surgeon Dissected Grafts
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eye Bank Pre-cut Grafts (N=20) | Surgeon Dissected Grafts (N=20)
graft dislocation and reattachment (Eye disorders) | 2 (2) | 2 (2)
graft rejection episode (Eye disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No